CLINICAL TRIAL: NCT03103620
Title: Safety And Effectiveness Evaluation Of COBRA PzF™ Coronary Stent System: A French Observational Postmarketing Registry
Brief Title: Safety and Effectiveness Evaluation of COBRA PzF Coronary Stent System: A Post Marketing Observational Registry
Acronym: eCOBRA
Status: Completed | Type: Observational
Sponsor: CeloNova BioSciences, Inc. (Industry)
Collaborators: AlpinARC (Unknown)
Responsible Party: Sponsor
Other Study IDs: COBRA 2013-01
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Stable Angina; Unstable Angina; ACS - Acute Coronary Syndrome; STEMI; NSTEMI - Non-ST Segment Elevation MI; Myocardial Infarction
MeSH Terms: conditions — Angina, Stable; Angina, Unstable; Acute Coronary Syndrome; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: COBRA PzF Coronary Stent System — COBRA PzF Coronary Stent System

SUMMARY:
A multi-center, prospective, consecutive enrolled, observational registry. The population being studied includes all patients undergoing treatment of "de novo" lesions in native coronary vessels, saphenous vein graft and/or arterial bypass conduits with the COBRA PzF coronary stent system. The registry will primarily assess the rate of MACE (cardiac death, myocardial infarction and clinically driven target lesion revascularization.

ELIGIBILITY:
Inclusion Criteria:

Patient has given oral consent to participate in the registry Patient is implanted with a COBRA PzF stent Target lesion(s) is/are "de novo"

Exclusion Criteria:

Pregnancy Age <18 years Refusal or inability to give oral consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing treatment of "de novo" lesions in native coronary vessels, saphenous vein graft and/or arterial bypass conduits with the COBRA PzF coronary stent system
Sampling Method: Non-Probability Sample
Enrollment: 1027 (Actual)
Dates: Start 2015-09-10 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
MACE | 12 months
  Composite clinical endpoint of cardiac death, myocardial infarction, and clinically driven target lesion revascularization

SECONDARY OUTCOMES:
Stent thrombosis | 12 months
  Stent thrombosis (according to ARC definition)
TVR and TLR | 12 months
  Target vessel and lesion revascularization
DAPT | 12 months
  Mean length of dual antiplatelet therapy

CONTACTS AND LOCATIONS:
Overall Officials: Luc Maillard, MD, Principal Investigator — Clinique Axium
Locations (18):
- France (18):
  - Clinique Axium, Aix
  - GCS Cardio, Annecy
  - SCM Angioscan, Antony
  - Clinique La Casamance, Aubagne
  - Centre Hospitalier, Avignon
  - Clinique La Fourcade, Bayonne
  - Centre Hospitalier, Brivé
  - Clinique des Domes, Clermont
  - Clinique Cardiologie, Évecquemont
  - Clinique Mutualiste, Grenoble
  - Centre Hospitalier, Haguenau
  - Infirmerie Protestante, Lyon
  - Clinique du Pont de Chaume, Montauban
  - Clinique du Millenaire, Montpellier
  - Centre Hospitalier, Pau
  - Clinique St-Martin, Pessac
  - Polyclinique de Courlancy, Reims
  - Clinique St Hilaire, Rouen

IPD SHARING:
Plan to Share IPD: No